CLINICAL TRIAL: NCT01264965
Title: Opioids Versus Extra Strength Acetaminophen for the Management of Moderate Persistent Non-cancer Pain
Brief Title: Non-cancer Pain and Cognitive Impairment: A Disabling Relationship
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment problems
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-238-B
Record Dates: First submitted 2010-12-20; First posted 2010-12-22 (Estimated); Results first posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-11

CONDITIONS: Arthritis; Pain; Cognitive Impairment
Keywords: Pain; Analgesia; Cognitive impairment; Randomized controlled trial; Physical function
MeSH Terms: conditions — Arthritis; Pain; Cognitive Dysfunction; Agnosia | interventions — acetaminophen, aspirin, caffeine drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetaminophen (Active Comparator)
  Interventions: Drug: extra strength acetaminophen
- Long Acting Oxycodone (Active Comparator)
  Interventions: Drug: long acting oxycodone

INTERVENTIONS:
Drug: long acting oxycodone — 10mg twice daily
  Arms: Long Acting Oxycodone
Drug: extra strength acetaminophen — 1,000 mg twice daily
  Arms: Acetaminophen

SUMMARY:
To compare the efficacy of long-acting oxycodone to extended-release acetaminophen in older persons with no and mild to moderate cognitive impairment and persistent moderate or higher intensity non-cancer lower extremity arthritis pain; and Describe the association of change in non-cancer pain self-report with an older adults functional status (BPI and WOMAC and brief physical performance measure) and to determine if cognitive status modifies this relationship.

ELIGIBILITY:
Inclusion Criteria:

1. age over 65
2. Pain at least 3 months duration
3. Pain greater in lower extremity than other anatomical site with ambulation
4. Pain self-report of moderate intensity of higher on an average day
5. Community-dwelling
6. Ambulatory
7. Physician states participants have decision-making capacity to enroll into the trial
8. Participants with cognitive impairment have a reliable caregiver
9. Inadequate pain relief from NSAIDS and/or acetaminophen in the past

Exclusion Criteria:

1. Current cancer requiring chemotherapy
2. History of addiction to opioids or other controlled substance
3. Consumes more than 2 alcoholic drinks a day
4. Severe balance disturbance
5. Intra-articular steroid injection in the past 6 weeks

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago Medical Center Outpatient Senior Health Center South Shore, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Enrolled Patients: This study was initially designed as a randomized crossover trial comparing extra strength acetaminophen (1,000 mg twice daily) to long acting oxycodone (10 mg twice daily). Unfortunately the treatment group assignments were lost and therefore there is no information on which treatment sequence patients were assigned to.
Period: Overall Study
Arm/Group | All Enrolled Patients
Started | 25
Completed | 15
Not Completed | 10
Not completed — Withdrawal by Subject | 10

BASELINE CHARACTERISTICS:
Arm/Group | All Enrolled Patients
Number analyzed (Participants) | 25
Age, Continuous [Mean (Full Range); unit: years] | 79.4 [67 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Pain Self-report on the Brief Pain Inventory and WOMAC
Time Frame: 14 days
Population: No data are available for this outcome (study records were lost).
Arm/Group | All Enrolled Patients
Number analyzed (Participants) | 0

2. Secondary Outcome: Discontinuation of Study Drug, Short Physical Performance Battery
Time Frame: 14 days
Population: No data are available for this outcome (study records were lost).
Arm/Group | All Enrolled Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: This study was initially designed as a randomized crossover trial comparing extra strength acetaminophen (1,000 mg twice daily) to long acting oxycodone (10 mg twice daily). Unfortunately the treatment group assignments were lost and therefore there is no information on which treatment sequence patients were assigned to. In addition, no information is available on the timing of adverse events. As a result, adverse events can only be reported for the entire group of enrolled patients.
Arm/Group | All Enrolled Patients
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 10/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Enrolled Patients (N=25)
Nausea (Gastrointestinal disorders) | 9
Confusion (Psychiatric disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No